CLINICAL TRIAL: NCT05070416
Title: Clinical Evaluation of Lithium Disilicate CAD/CAM Crowns
Brief Title: Lithium Disilicate Crowns Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Material did not perform accordingly in other clinical trials.
Sponsor: Ivoclar Vivadent AG (Industry)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LL3986001; HUM00191892 (Registry Identifier: IRBMED (Medical School Institutional Review Board))
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-09

CONDITIONS: Caries; Dental Trauma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Crowns self-adhesively cemented (Experimental): Group 1 receives crowns with an occlusal thickness of 1.5 mm and luted with a self-adhesive, self-curing resin cement (SpeedCem Plus, Ivoclar Vivadent AG).
  Interventions: Device: Lithium disilicate crowns
- Crowns adhesively luted (Experimental): Group 2 receives crowns with an occlusal thickness of 1.2 mm delivered with a dual-curing resin cement (Variolink Esthetic (DC),Ivoclar Vivadent AG).
  Interventions: Device: Lithium disilicate crowns

INTERVENTIONS:
Device: Lithium disilicate crowns — The study population is separated in two groups. The teeth will be etched in total etch mode with 37% phosphoric acid (Total Etch, Ivoclar Vivadent AG). After the application of Adhese Universal-adhesive (Ivoclar Vivadent AG), MultiCore Flow (Ivoclar Vivadent AG) will be applied. The crowns will be polished, then etched with IPS Ceramic Etching Gel (Ivoclar Vivadent AG) and conditioned with Monobond Plus (Ivoclar Vivadent AG). The crowns will be luted as described for group 1 or 2. A final intraoral polishing step will be done with OptraGloss (Ivoclar Vivadent AG). All required light-curing steps are conducted with Bluephase G4 (Ivoclar Vivadent AG).

SUMMARY:
CAD-CAM crowns made of experimental lithium disilicate (shades A1, A2 and A3) are placed in patients by using either a dual-curing adhesive or a self-adhesive luting material in combination with total etch/universal bonding agent.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be at least 18 years of age, of either gender, and of any ethnic background.
* Each patient should have at least one carious lesion or defective restoration to be restored on a maxillary or mandibular premolar or molar tooth.
* Each lesion or defective restoration should exhibit sufficient size or loss of tooth structure requiring a full crown restoration.
* The tooth should have at least one opposing tooth in occlusion and one adjacent tooth with an intact proximal contact.
* All teeth will test vital and be asymptomatic at the beginning of treatment. No more than two restorations will be placed per patient.

Exclusion Criteria:

* Devital or sensitive teeth
* Teeth with prior endodontic treatment of any kind
* Teeth with a history of direct or indirect pulp capping procedures
* Patients with significant untreated dental disease to include periodontitis and/or rampant caries
* Women who self-report that they are possibly pregnant, pregnant, or lactating, as elective dental treatment is not indicated at these times
* Patients with a self-reported past history of allergies to the materials to be used in the study including composite resin cements or ceramic restorative materials
* Patients unable to return for the recall appointments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis J. Fasbinder, DDS, Principal Investigator — University of Michigan School of Dentistry, Department of Cariology, Restorative Sciences & Endodontics
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 04.10.2021 to 01.03.2023 in the clinic.
Units Other Than Participants: crowns
Period: Overall Study
Arm/Group | Crowns self-adhesively cemented | Crowns adhesively luted
Started | 3; 3 crowns | 5; 5 crowns
Completed | 3; 3 crowns | 5; 5 crowns
Not Completed | 0; 0 crowns | 0; 0 crowns

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Crowns self-adhesively cemented | Crowns adhesively luted | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Customized [Number; unit: participants]
  > 18 years | 3 | 5 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 5 | 5
  Male | 3 | 0 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Crowns With Short-term Post-operative Sensitivity
Description: assessed by patient's weekly feedback for 4 weeks after the treatment rating sensitivity from 1 "no sensitivity" to 4 "severe discomfort noted routinely with cold or pressure stimulation"
Time Frame: 4 weeks
Measure: Number; unit: Crowns
Units Other Than Participants: Crowns
Arm/Group | Crowns self-adhesively cemented | Crowns adhesively luted
Number analyzed (Participants) | 3 | 5
Number analyzed (Crowns) | 3 | 5
Crowns | 0 | 0

2. Secondary Outcome: Quality Criteria (Modified FDI Criteria)
Description: assessed following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable" (e.g. surface lustre, Staining, and colour match of restorations)
Time Frame: 4 weeks
Population: The clinical trial was early terminated and therefore, only the quality criteria of some participants could be assessed in detail.
Measure: Number; unit: Crowns
Units Other Than Participants: Crowns
Arm/Group | Crowns self-adhesively cemented | Crowns adhesively luted
Number analyzed (Participants) | 3 | 5
Number analyzed (Crowns) | 3 | 5
Crowns
  FDI 1 Surface Luster, FDI Score 1 | 3 | 5
  FDI 1 Surface Luster, FDI Score 2-5 | 0 | 0
  FDI 2 Surface Staining, FDI Score 1 | 3 | 5
  FDI 2 Surface Staining, FDI Score 2-5 | 0 | 0
  FDI 3 Colour, FDI Score 1 | 2 | 5
  FDI 3 Colour, FDI Score 2 | 1 | 0
  FDI 3 Colour, FDI Score 3-5 | 0 | 0
  FDI 6 Marginal Adaption, FDI Score 1 | 3 | 5
  FDI 6 Marginal Adaption, FDI Score 2-5 | 0 | 0
  FDI 8 Approximal anatomical form, FDI Score 1 | 3 | 5
  FDI 8 Approximal anatomical form, FDI Score 2-5 | 0 | 0
  FDI 10 Patient view, FDI Score 1 | 3 | 5
  FDI 10 Patient view, FDI Score 2-5 | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Crowns self-adhesively cemented | Crowns adhesively luted
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 0/3 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/16/NCT05070416/Prot_SAP_002.pdf